CLINICAL TRIAL: NCT07359781
Title: Assessment of Exercise Motivation in Adolescent Idiopathic Scoliosis: Validity and Reliability Study of the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2)
Brief Title: Validity and Reliability of the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) in Adolescents With Idiopathic Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Hafize Hilal KARGIN, Lecturer, Nigde Omer Halisdemir University
Other Study IDs: OHU-HHK-QV-2026-01
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Adolescence Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis, Exercise motivation, Behavioral regulation, Validity and reliability, Self-determination theory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents With Idiopathic Scoliosis: Adolescents aged 10-19 years diagnosed with adolescent idiopathic scoliosis who have been receiving scoliosis-specific exercise therapy for at least two months and who voluntarily participate in the study.
  Interventions: Other: Questionnaire Assessment

INTERVENTIONS:
Other: Questionnaire Assessment — No intervention is administered. Participants complete self-reported questionnaires (BREQ-2, QPSSE motivation subscale, and EMI-2) for the assessment of exercise motivation.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a spinal condition that develops during adolescence and often requires long-term conservative treatment, including scoliosis-specific therapeutic exercises. The success of exercise-based treatment largely depends on adolescents' motivation to start and continue exercising. However, exercise motivation has not been adequately evaluated in adolescents with idiopathic scoliosis using validated tools specific to this population.

The Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) is a widely used questionnaire based on Self-Determination Theory that assesses different types of motivation toward exercise. Although the Turkish version of the BREQ-2 exists, its validity and reliability have not yet been examined in adolescents with idiopathic scoliosis.

The purpose of this study is to evaluate the validity and reliability of the Turkish version of the BREQ-2 in adolescents diagnosed with idiopathic scoliosis. Adolescents aged 10-19 years who have been participating in scoliosis-specific therapeutic exercise programs for at least two months will be invited to complete online questionnaires. The results of this study will help determine whether the BREQ-2 is an appropriate tool for assessing exercise motivation in this population and may support the development of individualized motivational strategies in scoliosis rehabilitation.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformity of the spine that emerges during growth and often requires prolonged conservative management. Physiotherapeutic scoliosis-specific exercises (PSSE) are recommended in international guidelines and have demonstrated effectiveness in controlling curve progression and improving functional outcomes. However, adherence to exercise programs remains a major challenge, particularly during adolescence, where motivation plays a critical role in sustaining health-related behaviors.

Exercise motivation is commonly conceptualized within the framework of Self-Determination Theory as a continuum ranging from amotivation to intrinsic motivation. The Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) is a theory-based, multidimensional instrument designed to assess motivational regulation underlying exercise behavior. While the BREQ-2 has demonstrated strong psychometric properties across different populations, its validity and reliability have not been established in adolescents with idiopathic scoliosis.

This study is designed as a methodological, cross-sectional validation study aiming to evaluate the validity, reliability, and applicability of the Turkish version of the BREQ-2 in adolescents with idiopathic scoliosis. Participants aged 10-19 years who have been receiving scoliosis-specific therapeutic exercise treatment for at least two months will be recruited. Data will be collected using online questionnaires, including the BREQ-2, the motivation subscale of the Questionnaire on Physiotherapeutic Scoliosis-Specific Exercises (QPSSE), and the Exercise Motivations Inventory-2 (EMI-2).

Internal consistency of the BREQ-2 will be assessed using Cronbach's alpha coefficients. Test-retest reliability will be evaluated using the intraclass correlation coefficient (ICC) with a two-week interval between administrations. Criterion-related validity will be examined by analyzing correlations between BREQ-2 scores and scores obtained from the QPSSE motivation subscale and the EMI-2. Statistical analyses will be performed using appropriate correlation methods based on data distribution.

The findings of this study are expected to provide evidence regarding the psychometric adequacy of the BREQ-2 for assessing exercise motivation in adolescents with idiopathic scoliosis. Establishing a valid and reliable motivation assessment tool may contribute to improved evaluation of treatment adherence and support the development of individualized motivational approaches in scoliosis rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 and 19 years
* Diagnosed with adolescent idiopathic scoliosis
* Receiving scoliosis-specific therapeutic exercise treatment for at least 2 months
* Able to read and write in Turkish
* Volunteered to participate in the study and provided informed consent

Exclusion Criteria:

* Presence of congenital or neuromuscular scoliosis
* Presence of systemic disease
* Presence of syndromic conditions such as Marfan syndrome or Ehlers-Danlos syndrome

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of adolescents aged 10 to 19 years who have been diagnosed with adolescent idiopathic scoliosis and are currently receiving scoliosis-specific exercise-based physiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) | Baseline assessment; test-retest reliability assessed over a 2-week interval
  The primary outcome is the psychometric evaluation of the Turkish version of the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) in adolescents with idiopathic scoliosis, including internal consistency, test-retest reliability, and criterion-related validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) sharing has not yet been determined. Decisions regarding data sharing will be made following completion of the study, in accordance with institutional policies, ethical approval conditions, and data protection regulations.